CLINICAL TRIAL: NCT04158830
Title: A Pragmatic Randomized Study Comparing 81 mg Aspirin Versus 162 mg Aspirin in the Prevention of Preeclampsia During Pregnancy
Brief Title: Aspirin (ASA) Therapy and Preeclampsia Prevention
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI is no longer at this University.
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 19-06959-FB
Record Dates: First submitted 2019-10-18; First posted 2019-11-12 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Preeclampsia
Keywords: prevention; aspirin therapy
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in consecutive order, entering their basic information (name, date of birth, medical record number, date/time of randomization, randomization number) on a master log.
  Group 1- (total of up to 450 subjects) designated by odd numbers in the randomization pattern [1-001, 1-003, 1-005, etc. to 899] oral dose: 81 mg aspirin daily: Rx 81 mg ASA, 1 tablet daily (1 bottle of 200 tablets/patient)
  Group 2-(total of up to 450 subjects) designated by even numbers in the randomization pattern [2-002, 2-004, 2-006, etc. to 900] oral dose: 162 mg aspirin daily: Rx 81 mg ASA, 2 tablets daily (1 bottle of 400 tablets/patient)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - ACOG recommended dose (Other): oral dose: 81 mg aspirin daily; designated by odd number assignment [1-001, 1-003, 1-005, etc. to 899]
  Interventions: Drug: Aspirin 81 mg Enteric Coated Tab - 1 tablet
- Group 2 - Comparison Dose (Active Comparator): oral dose: 162 mg aspirin daily; designated by even number assignment [2-002, 2-004, 2-006, etc. to 900]
  Interventions: Drug: Aspirin 81 mg Enteric Coated Tab - 2 tablets

INTERVENTIONS:
Drug: Aspirin 81 mg Enteric Coated Tab - 1 tablet — take one (1) 81 mg tablet each evening
  Other Names: Group 1 - ACOG recommended dose
  Arms: Group 1 - ACOG recommended dose
Drug: Aspirin 81 mg Enteric Coated Tab - 2 tablets — take two (2) 81 mg tablets each evening
  Other Names: Group 2 - Comparison Dose
  Arms: Group 2 - Comparison Dose

SUMMARY:
According to U.S. Pharmacist® "low-dose aspirin refers to dosages between 81 mg and 325 mg taken every day to prevent heart attacks, strokes, and colon cancer." It has been found through research that low-dose aspirin also decreases the risk of preeclampsia. The American College of Obstetrics and Gynecologists (ACOG) recommends low-dose aspirin (81mg/day) for women at high risk of preeclampsia. However, some researchers report that a dose of aspirin < 100 mg/day does not seem to decrease the risk of preeclampsia. Another trial studying patients who are at a high risk for preterm preeclampsia, reported a reduction in the occurrence of preeclampsia among patients taking aspirin at a dose of 150 mg.

The purpose of this pragmatic randomized study is to compare the difference in the effectiveness of two doses of aspirin: 81 mg versus 162 mg in the prevention of preeclampsia in pregnant women who are at a moderate to high risk for developing preeclampsia.

DETAILED DESCRIPTION:
Rationale - The risk factors associated with preeclampsia (early-onset and late-onset, singleton deliveries) include the following maternal characteristics and clinical factors (Washington State, 2003-2008; ACOG 2018): age < 20 years, age >34 years, African-American race, marital status-single, first pregnancy, diabetes mellitus, chronic hypertension, infertility treatment, infant sex male, and congenital anomalies.

Low dose aspirin decreases the risk of preeclampsia. The 2018 ACOG Committee Opinion on "Low-dose aspirin use during pregnancy" recommends the use of 81mg/day of aspirin for patients with risk factors for preeclampsia. However, it has been reported that a dose of aspirin < 100 mg/day does not seem to decrease the risk of preeclampsia.

Rolnick et al., studying patients at high risk for preterm preeclampsia, reported a 63% relative risk reduction among patients taking aspirin at 150mg per day versus placebo. We anticipate a more conservative rate of 40% relative risk reduction, from 35% to 21%, for patients taking 162mg per day.

Study/Project Population - We will include pregnant women up to 28.0 weeks gestation coming to the Regional One Health Obstetric (OB) Clinic for prenatal care, who meet ACOG's definition of high or moderate risk of developing preeclampsia during their current pregnancy (Low risk subjects will not be included).

Those risk factors are:

High Rish [ACOG recommends low-dose aspirin if the patient has one or more of these high-risk factors.]

1. History of preeclampsia, especially when accompanied by an adverse outcome
2. Multifetal gestation
3. Chronic hypertension
4. Type 1 or 2 Diabetes mellitus
5. Renal disease [>300 mg/24-hour urine; protein creatinine ratio > 0.3; 1+ proteinuria; creatinine >1.2]
6. Autoimmune disease (for example, systemic lupus erythematosus, antiphospholipid syndrome)

   Moderate Risk [ACOG recommends consideration of low-dose aspirin if the patient has more than one of these moderate-risk factors. Moderate-risk factors vary in their association with increased risk of preeclampsia.]
7. Nulliparity
8. Obesity (body mass index greater than 30)
9. Family history of preeclampsia (mother or sister)
10. Sociodemographic characteristics (African American race, low socioeconomic status)
11. Age 35 years or older
12. Personal history factors (e.g., low birthweight or small for gestational age, previous adverse pregnancy outcome, more than 10-year pregnancy interval)

    Low Risk [ACOG does not recommend low-dose aspirin.]
13. Previous uncomplicated full-term delivery

Research Design - This is a prospective clinical trial with binomial outcome and random assignment to two independent study groups, with a 1:1 ratio of assignment to 162mg versus 81mg of aspirin recommended daily.

For our sample size calculation, we use a one-sided Likelihood Ratio Chi-square Test for two proportions, with a Type I error rate of 5%, and power of 80%. To detect a 40% relative risk reduction in term preeclampsia prevalence, from 15% to 9%, requires a total (N)umber of 720 patients. We estimate a 20% attrition due to causes including non-compliance, delivering at other hospitals, and non-hospital deliver; and therefore, plan to recruit 900 patients (450 patients per group).

To compare the ratios of preeclampsia incidence between two assigned groups, assigned to 162mg or 81mg of daily aspirin, we plan to use a Likelihood Ratio Chi-square Test or Fisher's exact test.

We anticipate a 12-month recruitment period for this study. The number of deliveries at Regional One Health (ROH) for the years 2017 and 2018 were 3325 and 3031 respectively. However, for this same period, the number of patients receiving prenatal care through Regional One Health Outpatient Center (MedPlex) were 1564 and 1651 respectively. This reveals that approximately 50% of those patients delivering at ROH did not receive prenatal care through Regional One Health.

Study/Project Procedures - We will screen for eligibility by reviewing the clinic appointment lists, matching patient's reason for visit with key words indicating they are likely candidates. Subjects meeting inclusion criteria will be further screened for eligibility during their OB clinic visit. The willing subjects will have the informed consent presented, thoroughly explained, and given an opportunity to ask questions.

Consented subjects will be randomly assigned and prescribed a daily dosage of 81 mg or 162 mg of aspirin to be taken each evening at bedtime. (See additional description below). Study drug bottles will be dispensed on the day of enrollment. Subjects will be instructed to continue taking the aspirin according to their randomization through the end of their pregnancy.

Subjects will be randomized in consecutive order, entering their basic information (name, date of birth, medical record number, date/time of randomization, randomization number) on a master log.

Patients recruited in the study will undergo a standard treatment ultrasound during the first trimester. At the time of consent, study subjects will be asked about their willingness to have a maternal uterine artery doppler ultrasound performed specifically for research. The maternal uterine artery doppler ultrasound will require an additional 3 minutes of the subject's time. If the subject agrees to participate in this portion of the study, they will initial the affirmative response line of the consent form.

The additional information collected during the maternal uterine artery doppler ultrasound will add to the body of knowledge used as predictors of preeclampsia. This information will not be used for clinical management.

We will collect data from the patient's electronic medical record (EMR) and the patient's fetus'/newborn's EMR, established at Regional One Health (clinic and hospital). This will include information pertaining to health history, current medical treatment, medications, pregnancy ultrasound scans, labor, delivery, and birth information.

Collected paper records will be maintained in the research office under locked conditions. Electronic data will be retrieved, entered and stored in a study titled REDCap Data File, utilizing password protection for access. We will request the guidance and assistance of the Center for Biomedical Informatics (CBMI) personnel as is needed.

Outcome Measures - Our primary outcome will be the occurrence of preeclampsia. Preeclampsia will be defined according to the 2018 American College of Obstetricians and Gynecologists recommendations.

Interim analysis will be conducted after 318 enrolled subjects have delivered, evaluating the outcomes of: 'no preeclampsia,' 'preterm preeclampsia,' and 'term preeclampsia.' Enrollment will continue if the results of the first interim analysis are inconclusive. At that time, continuation of enrollment to 646 subjects delivered with a second interim analysis, or up to enrollment of 900 subjects delivered for a third, final analysis.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females ages 14 to 50 years old
* Up to 28.0 weeks gestation (may initially base on last menstrual period (LMP), but confirmed with ultrasound (US)
* Be at high risk or moderate risk for developing preeclampsia as defined by the American College of Obstetrics and Gynecologists (ACOG-2018), the Society for Maternal-Fetal Medicine (SMFM-2018), and the United States Preventive Services Task Force (USPSTF-2017)

Exclusion Criteria:

* Less than 14 years old or greater than 50 years old
* Allergy or contraindication to taking aspirin (i.e. nasal polyps, asthma with aspirin-induced bronchoconstriction)
* History of gastrointestinal bleeding
* Active peptic ulcer disease
* Other sources of active Gastrointestinal/Genitourinary bleeding
* Physician or provider refusal
* Patient refusal
* History of bleeding or clotting disorder (i.e. Factor V, von Willebrand, hemophilia)
* Severe renal failure (Glomerular Filtration Rate < 10 ml/min)
* Taking aspirin prior to pregnancy

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women only
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Preeclampsia | approximately 30 weeks; from 12 weeks gestation until the day of delivery
  Occurrence of preeclampsia: categorized as - none, preterm, or term

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Mari, MD, FACOG, Principal Investigator — OB/ GYN Department Professor and Chair
Locations (1):
- Regional One Health, Obstetrics Outpatient Clinic, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roberge S, Bujold E, Nicolaides KH. Aspirin for the prevention of preterm and term preeclampsia: systematic review and metaanalysis. Am J Obstet Gynecol. 2018 Mar;218(3):287-293.e1. doi: 10.1016/j.ajog.2017.11.561. Epub 2017 Nov 11. PMID 29138036
- [Result] ACOG Committee Opinion No. 743: Low-Dose Aspirin Use During Pregnancy. Obstet Gynecol. 2018 Jul;132(1):e44-e52. doi: 10.1097/AOG.0000000000002708. PMID 29939940
- [Result] Lisonkova S, Joseph KS. Incidence of preeclampsia: risk factors and outcomes associated with early- versus late-onset disease. Am J Obstet Gynecol. 2013 Dec;209(6):544.e1-544.e12. doi: 10.1016/j.ajog.2013.08.019. Epub 2013 Aug 22. PMID 23973398
- [Result] Roberge S, Nicolaides K, Demers S, Hyett J, Chaillet N, Bujold E. The role of aspirin dose on the prevention of preeclampsia and fetal growth restriction: systematic review and meta-analysis. Am J Obstet Gynecol. 2017 Feb;216(2):110-120.e6. doi: 10.1016/j.ajog.2016.09.076. Epub 2016 Sep 15. PMID 27640943
- [Result] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Result] Seidler AL, Askie L, Ray JG. Optimal aspirin dosing for preeclampsia prevention. Am J Obstet Gynecol. 2018 Jul;219(1):117-118. doi: 10.1016/j.ajog.2018.03.018. Epub 2018 Mar 26. No abstract available. PMID 29588190
- [Result] LeFevre ML; U.S. Preventive Services Task Force. Low-dose aspirin use for the prevention of morbidity and mortality from preeclampsia: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2014 Dec 2;161(11):819-26. doi: 10.7326/M14-1884. PMID 25200125
- [Result] Lovgren TR, Dugoff L, Galan HL. Uterine artery Doppler and prediction of preeclampsia. Clin Obstet Gynecol. 2010 Dec;53(4):888-98. doi: 10.1097/GRF.0b013e3181fbb687. PMID 21048456